CLINICAL TRIAL: NCT03371732
Title: Effectiveness of Screening and Brief Interventions for Alcohol and/or Tobacco During Breast Cancer Treatment: A Phase III, Pilot Prospective Randomized Trial (ONKODETOX)
Brief Title: Effectiveness of Screening and Brief Interventions for Alcohol and Tobacco During Breast Cancer Treatment (ONKODETOX)
Acronym: ONKODETOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IB2013-ONKODETOX
Record Dates: First submitted 2017-11-09; First posted 2017-12-13 (Actual); Results first posted 2021-05-03 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer; Psychology, Social
Keywords: Psychological intervention Alcohol; Tobacco consumption; Substance use; Health risk behavior; Oncology setting; Women; Supportive care
MeSH Terms: conditions — Breast Neoplasms; Tobacco Use; Substance-Related Disorders; Health Risk Behaviors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Groupe 1 (Other): G1 : Motivational Intervention group
  Interventions: Behavioral: Motivational Intervention group
- Groupe 2 (Other): G2 : Educational advises group
  Interventions: Behavioral: Educational advises group

INTERVENTIONS:
Behavioral: Motivational Intervention group — Participants in the intervention group a one-session brief motivational intervention administered by a psychologist. This intervention consist in a single adapted motivational interview lasting 20-30 minutes, based on the principles of the trans-theoretical model and on the manual for motivational therapy. It is carried out by the same psychologist, trained and supervised for this type of intervention.
  Arms: Groupe 1
Behavioral: Educational advises group — Participants in this group benefit of brief educational advises (10 minutes interview maximum ; only on alcohol/tobacco consumption consequences on health), and received a pamphlet on the health effects of alcohol and tobacco consumption.
  Arms: Groupe 2

SUMMARY:
Despite scientific, clinical and political incentives, alcohol and/or tobacco screening and brief intervention (SBI) services are poorly implemented in oncology settings. Motivational brief interventions are recognized as particularly effective in changing health behaviors, especially consumption behaviors. The motivational approach is more and more used in primary care setting but still few studies explore its effectiveness with breast cancer patients.

This study aims to compare two intervention arms : educational advices intervention (EAI) versus brief motivational intervention (BMI) for alcohol and/or tobacco consumption in breast cancer women, during their treatment.

In this pilot prospective randomized trial, various psychological and behavioral, variables are measured (alcohol and tobacco consumption, distress, anxiety and depressive disorders, quality of life, motivation for change, empowerment) before the brief intervention, and after 3 and 6 month.

DETAILED DESCRIPTION:
Context :

It is now well documented that alcohol and tobacco reduce the effectiveness of a treatment, increase the side effects, favor the recurrence and/or secondary cancers and affects the quality of life of patients treated for cancer, including breast cancer. The announcement of the disease could create a window of opportunity for change in lifestyle for patients. The 2014-2019 French Cancer Plan emphasizes the need for the implementation of prevention and risk reduction related to alcohol and tobacco. A screening, brief motivational and referral to treatment program, specifically dedicated to oncology can be public health approach aiming to reduce the harmful consequences of substance misuse and improving the prognosis and quality of life of consumers at risk.

Main objective :

Evaluate effectiveness of a brief motivational intervention for alcohol and/or tobacco in short (3 month) and medium (6 month) terms in breast cancer patients, in a prospective randomized pilot study.

Secondary objectives :

* Determine the behavioral and psychopathological specific characteristics of the patient linked to change process and maintain.
* Define a brief intervention for alcohol/tobacco consumption model adapted and integrated to patient treated for cancer according to psychosocial factors highlighted.

The investigators will seek to highlight the benefit of a motivational brief intervention versus standardized educational advice. The specificity of these interventions is to be integrated in an interview integrating a systematic screening of the emotional distress of the patient, of these concerns as well as of his perceived need for aids.

Method :

This is a randomized clinical trial comparing two interventions. The trial includes 200 primary breast cancer patients with a positive AUDIT-C score and/or are tobacco consumers, randomly placed in two groups :

G1 : Motivational Intervention group (N = 100) : Participants in the intervention group benefit a one-session brief motivational intervention administered by a psychologist. This intervention consist in a single adapted motivational interview lasting 20-30 minutes, based on the principles of the trans-theoretical model and on the manual for motivational therapy. It is carried out by the same psychologist, trained and supervised for this type of intervention.

G2 : Educational advises group (N = 100) : Participants in this group benefit of brief educational advises (10 minutes interview maximum), and received a pamphlet on the health effects of alcohol and tobacco consumption. For obvious ethical reasons, the investigators selected an intervention in the form of advice concerning the effects of the product and the submission of specific documentation (criteria not retained in the context of the brief intervention model). It did not seem possible to evaluate patients without offering them the possibility of a low threshold intervention.

Detailed scripts for each modality of intervention are realized.

Measurement :

Three sets of measurements are taken at baseline, 3-month and 6 month follow-up.

Primary Outcome measures: Clinically significant reduction (beneficial to health) of risk behaviours (alcohol and/or tobacco consumption) :

* Concerning subjects with only alcohol consumption at baseline : The intervention will be considered effective at 3 months if an individual decrease of 20% in the AUDIT score is observed at 3 months compared to the value collected at baseline; The intervention will be considered effective at 6 months if this 20% reduction is maintained at 6 months, still in relation to the value collected at baseline.
* The same applies to subjects with only tobacco consumption at baseline: The intervention will be considered effective at 3 months if an individual decrease of 20% in the number of cigarettes consumed per day is observed at 3 months compared to the value collected at baseline; The intervention will be judged effective at 6 months if this 20% reduction is maintained at 6 months, still in relation to the value collected at baseline.
* Finally, with regard to women with both alcohol and tobacco use at baseline :

The intervention will be considered effective if at least one of the two scores (AUDIT or number of cigarettes consumed per day) has decreased by 20% at 3 months (maintained at 6 months) compared to the value collected at baseline, with no increase in the other score.

Secondary outcome measures :

* Individual reduction of around 20% in average daily consumption of alcohol and/or tobacco (calculated on the basis of patients' consumption schedules) between inclusion and the first follow-up at 3 months, and maintenance of this success at the second follow-up at 6 months (with no increase in other consumption if the subject has both alcohol and tobacco consumption at inclusion);
* Description of the variables relating to the consumption of alcohol, tobacco, the current medico-psychological situation, psychological distress, anxio-depressive symptomatology, willingness to change alcohol and/or tobacco consumption habits;
* Improved quality of life in the experimental intervention arm compared to the standard intervention arm

Study procedure :

SCREENING-PRE-INCLUSION: Screening of distress and alcohol/tobacco consumptions is realized when the patients arrive in the oncology department for their chemotherapy treatment, by a research assistant-psychologist. Researchers propose to eligible patients to participate to the study. This first contact permits to check the absence of non-inclusion criteria; to ensure the informed consent of the person (an information and consent note will be given to him) and according to these elements, to define the provisional timetable for participation in the research.

T0 - INCLUSION AND RANDOMIZATION The research assistant retrieves the signed consent, ensuring a time available to return if necessary and carries out the research interview/assessment. The randomization is realized following this interview.

INTERVENTION: Brief intervention (G1 : Brief motivational intervention or G2 : educational advices) are conducted by the research assistant-psychologist, at the Institut Bergonié or by telephone if needed.

T1: MONITORING - FOLLOW-UP(3 months) Assessments are repeated, when the patient comes at the Institut Bergonié, by telephone if necessary.

T2: MONITORING - FOLLOW-UP (6 months) Assessments are repeated, when the patient comes at the Institut Bergonié, by telephone if necessary.

Randomization procedure :

The randomization procedure is done via the TENALEA server, managed by the Epidemiological and Clinical Research Unit (UREC) of the Bergonié Institute.

Expected results :

Highlighting:

* The efficacy of motivational brief intervention on alcohol and tobacco consumption in patients treated for breast cancer ; versus educational advices intervention.
* Psychosocial risk factors involved in maintaining problematic consumption or in the rapid relapse of tobacco/alcohol consumption.

ELIGIBILITY:
Inclusion Criteria :

* women with primary breast cancer, without ongoing support for substance use.
* An AUDIT-C score >1 or more than one cigarette smoked per day.
* Individuals able to consent to benefit of intervention focused on substance use. (Karnofsky Index >70).

Exclusion Criteria :

* Patients who currently use substances for which a second-line care is already committed.
* Patients with a Karnofsky index <70.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marion BARRAULT-COUCHOURON, PhD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonie, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Arm 1: Motivational Intervention group
  Motivational Intervention group: Participants in the intervention group a one-session brief motivational intervention administered by a psychologist. This intervention consist in a single adapted motivational interview lasting 20-30 minutes, based on the principles of the trans-theoretical model and on the manual for motivational therapy. It is carried out by the same psychologist, trained and supervised for this type of intervention.
- Arm 2: Arm 2: Educational advises group
  Educational advises group: Participants in this group benefit of brief educational advises (10 minutes interview maximum ; only on alcohol/tobacco consumption consequences on health), and received a pamphlet on the health effects of alcohol and tobacco consumption.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 51 | 53
Completed | 39 | 46
Not Completed | 12 | 7
Not completed — Withdrawal by Subject | 9 | 3
Not completed — Refusal to continue | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Arm 2: Arm 2 : Educational advises group
  Educational advises group: Participants in this group benefit of brief educational advises (10 minutes interview maximum ; only on alcohol/tobacco consumption consequences on health), and received a pamphlet on the health effects of alcohol and tobacco consumption.
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 51 | 53 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (10.4) | 48.0 (8.9) | 48.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 53 | 104
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Current family situation [Count of Participants; unit: Participants]
  Single | 4 | 6 | 10
  In a couple | 16 | 16 | 32
  Married | 21 | 25 | 46
  Divorced | 7 | 5 | 12
  Widowed | 3 | 1 | 4
Number of children [Mean (Standard Deviation); unit: Child] | 1.8 (0.9) | 1.8 (1.0) | 1.8 (1.0)
Level of education [Count of Participants; unit: Participants]
  No diploma | 2 | 1 | 3
  Below high school diploma | 10 | 10 | 20
  High school diploma to bachelor's degree (included) | 22 | 24 | 46
  Higher than bachelor's degree | 17 | 18 | 35
Profession [Count of Participants; unit: Participants]
  Farmer-operators | 0 | 0 | 0
  Artisans, merchants and company director | 0 | 2 | 2
  Company's exécutives and higher intellectual profession | 11 | 16 | 27
  Intermediate professions | 5 | 1 | 6
  Employees | 21 | 25 | 46
  Labor | 2 | 2 | 4
  Pensioners | 3 | 1 | 4
  Economically inactive | 9 | 6 | 15
Type of cancer [Count of Participants; unit: Participants]
  Canal carcinoma in situ | 0 | 4 | 4
  Ductal carcinoma infiltrant | 48 | 42 | 90
  Other | 3 | 7 | 10
Tumor extension stage [Count of Participants; unit: Participants] — Tumor extension T stage ranges from T0 (no primary tumor) to T4 (tumor invading an organ)
  Participants
    Missing | 4 | 3 | 7
    T0 | 1 | 2 | 3
    T1 | 9 | 11 | 20
    T2 | 23 | 21 | 44
    T3 | 13 | 13 | 26
    T4 | 1 | 3 | 4
Past treatment(s) [Count of Participants; unit: Participants]
  Surgery: No | 36 | 31 | 67
  Surgery: Yes | 15 | 22 | 37
  Chemotherapy: No | 22 | 27 | 49
  Chemotherapy: Yes | 29 | 26 | 55
  Radiotherapy: No | 49 | 50 | 99
  Radiotherapy: Yes | 2 | 3 | 5
  Hormonotherapy: No | 47 | 51 | 98
  Hormonotherapy: Yes | 4 | 2 | 6
  Without treatment: No | 41 | 38 | 79
  Without treatment: Yes | 10 | 15 | 25
Spouse's AUDIT-C score [Mean (Standard Deviation); unit: scores on a scale] — Alcohol Use Disorders IdentificationTest-Consumption (AUDIT-C) score ranges from 0 (No alcohol consumption) to 12 (alcohol dependence).Consumption profiles can be derived from this.
  Here the spouse's AUDIT-C score was presented.
  scores on a scale | 3.6 (2.6) | 3.4 (1.9) | 3.5 (2.2)
Currently, how many cigarettes per day do you smoke on average? [Mean (Standard Deviation); unit: Cigarettes per day] — Population: Among smokers only (N=54)
  Cigarettes per day
    number analyzed (Participants) | 27 | 27 | 54
    (all) | 11.5 (8.1) | 10.8 (6.9) | 11.1 (7.5)
Currently, how many cigarettes per day does the patient's spouse smoke on average? [Mean (Standard Deviation); unit: Cigarettes] — Population: For smokers only (N=54)
  Cigarettes
    number analyzed (Participants) | 27 | 27 | 54
    (all) | 11.5 (8.1) | 10.8 (6.9) | 11.1 (7.5)
In the past year, how often did the patient's spouse smoke? [Count of Participants; unit: Participants] — Population: Missing frequency = 23
  Participants
    number analyzed (Participants) | 39 | 42 | 81
    Never | 20 | 24 | 44
    At least once a week | 3 | 1 | 4
    Every day or almost every day | 16 | 17 | 33
DSM5 - Substance-related or addictive disorders (whole life) [Count of Participants; unit: Participants] — The Diagnostic and Statistical Manual of Mental Disorders, fifth edition, published by the American Psychiatric Association (APA) is a taxonomic and diagnostic tool.
  Participants
    No | 11 | 19 | 30
    Yes | 40 | 34 | 74
DSM5 - Substance-related or addictive disorders (whole life) [Count of Participants; unit: Participants] — The Diagnostic and Statistical Manual of Mental Disorders, fifth edition, published by the American Psychiatric Association (APA) is a taxonomic and diagnostic tool. Population: Only in patients with substance-related or addictive disorders (N=74)
  Participants
    Alcohol: number analyzed (Participants) | 40 | 34 | 74
    Alcohol: No | 36 | 34 | 70
    Alcohol: Yes | 4 | 0 | 4
    Tobacco: number analyzed (Participants) | 40 | 34 | 74
    Tobacco: No | 5 | 0 | 5
    Tobacco: Yes | 35 | 34 | 69
    Cannabis: number analyzed (Participants) | 40 | 34 | 74
    Cannabis: No | 39 | 34 | 73
    Cannabis: Yes | 1 | 0 | 1
    Other: number analyzed (Participants) | 40 | 34 | 74
    Other: No | 39 | 34 | 73
    Other: Yes | 1 | 0 | 1
DSM5 - Whole Life [Count of Participants; unit: Participants] — The Diagnostic and Statistical Manual of Mental Disorders, fifth edition, published by the American Psychiatric Association (APA) is a taxonomic and diagnostic tool.
  Participants
    Depressive disorders: No | 35 | 28 | 63
    Depressive disorders: Yes | 16 | 25 | 41
    Bipolar and related disorders: No | 51 | 51 | 102
    Bipolar and related disorders: Yes | 0 | 2 | 2
    Anxiety disorders: No | 38 | 39 | 77
    Anxiety disorders: Yes | 13 | 14 | 27
    OCD and related: No | 50 | 51 | 101
    OCD and related: Yes | 1 | 2 | 3
    Disorders related to trauma or stressors: No | 40 | 40 | 80
    Disorders related to trauma or stressors: Yes | 11 | 13 | 24
    Substance-related or Addictive: No | 11 | 19 | 30
    Substance-related or Addictive: Yes | 40 | 34 | 74
DSM5 - Substance-related or addictive disorders (current life) [Count of Participants; unit: Participants] — The Diagnostic and Statistical Manual of Mental Disorders, fifth edition, published by the American Psychiatric Association (APA) is a taxonomic and diagnostic tool.
  Participants
    No | 29 | 37 | 66
    Yes | 22 | 16 | 38
DSM5 - Current Life - Substance-related or addictive disorders [Count of Participants; unit: Participants] — Population: Only for patient with substance-related or addictive disorders (N=38)
  Participants
    Alcohol: number analyzed (Participants) | 22 | 16 | 38
    Alcohol: No | 19 | 15 | 34
    Alcohol: Yes | 3 | 1 | 4
    Tobacco: number analyzed (Participants) | 22 | 16 | 38
    Tobacco: No | 4 | 1 | 5
    Tobacco: Yes | 18 | 15 | 33
    Cannabis: number analyzed (Participants) | 22 | 16 | 38
    Cannabis: No | 21 | 16 | 37
    Cannabis: Yes | 1 | 0 | 1
    Other: number analyzed (Participants) | 22 | 16 | 38
    Other: No | 22 | 16 | 38
    Other: Yes | 0 | 0 | 0
DSM5 - Substance-related or addictive disorders (Current Life) [Count of Participants; unit: Participants] — The Diagnostic and Statistical Manual of Mental Disorders, fifth edition, published by the American Psychiatric Association (APA) is a taxonomic and diagnostic tool.
  Participants
    Depressive disorders: No | 47 | 48 | 95
    Depressive disorders: Yes | 4 | 5 | 9
    Depressive disorders: Missing | 0 | 0 | 0
    Bipolar and related disorders: No | 51 | 51 | 102
    Bipolar and related disorders: Yes | 0 | 2 | 2
    Bipolar and related disorders: Missing | 0 | 0 | 0
    Anxiety disorders: No | 45 | 43 | 88
    Anxiety disorders: Yes | 6 | 10 | 16
    Anxiety disorders: Missing | 0 | 0 | 0
    OCD and related: No | 50 | 52 | 102
    OCD and related: Yes | 0 | 1 | 1
    OCD and related: Missing | 1 | 0 | 1
    Disorders related to trauma or stressors: No | 47 | 50 | 97
    Disorders related to trauma or stressors: Yes | 3 | 3 | 6
    Disorders related to trauma or stressors: Missing | 1 | 0 | 1
Electronic cigarettes [Count of Participants; unit: Participants] — Population: Among smokers only (N=54)
  Participants
    number analyzed (Participants) | 27 | 27 | 54
    No | 25 | 24 | 49
    Yes | 2 | 3 | 5
Type of consumption of electronic cigarettes [Count of Participants; unit: Participants] — Population: Among electronic cigarette smokers only (N=5)
  Participants
    number analyzed (Participants) | 2 | 3 | 5
    With nicotine | 1 | 3 | 4
    Without nicotine | 1 | 0 | 1
Ongoing psychotropic treatment(s) [Count of Participants; unit: Participants]
  No | 35 | 35 | 70
  Yes | 16 | 18 | 34
Current monitoring with regard to behaviour/emotional state [Count of Participants; unit: Participants]
  Missing | 0 | 1 | 1
  No | 38 | 36 | 74
  Yes | 13 | 16 | 29
Type of professional [Count of Participants; unit: Participants] — Population: In patients with current monitoring of behaviour/emotional state (N=29)
  Participants
    Psychologist: number analyzed (Participants) | 13 | 16 | 29
    Psychologist: No | 3 | 3 | 6
    Psychologist: Yes | 10 | 13 | 23
    Psychiatrist: number analyzed (Participants) | 13 | 16 | 29
    Psychiatrist: No | 11 | 14 | 25
    Psychiatrist: Yes | 2 | 2 | 4
    Health professional specialising in tobaccoology and addiction: number analyzed (Participants) | 13 | 16 | 29
    Health professional specialising in tobaccoology and addiction: No | 13 | 15 | 28
    Health professional specialising in tobaccoology and addiction: Yes | 0 | 1 | 1
    Other professional: number analyzed (Participants) | 13 | 16 | 29
    Other professional: No | 12 | 16 | 28
    Other professional: Yes | 1 | 0 | 1
AUDIT Score (patient) [Mean (Standard Deviation); unit: scores on a scale] — Alcohol Use Disorders Identification Test-Consumption (AUDIT-C) score ranges from 0 (No alcohol consumption) to 12 (alcohol dependence). Consumption profiles can be derived from this.
  scores on a scale | 3.4 (4.2) | 2.9 (2.0) | 3.2 (3.3)
Score Audit categorical variable (Patient) [Count of Participants; unit: Participants] — Alcohol Use Disorders Identification Test-Consumption (AUDIT-C) score ranges from 0 (No alcohol consumption) to 12 (alcohol dependence). Consumption profiles can be derived from this
  Participants
    No consumption | 11 | 3 | 14
    Low-risk consumption | 33 | 44 | 77
    Harmful consumption | 3 | 6 | 9
    Probable dependency | 4 | 0 | 4
Fagerström score [Mean (Standard Deviation); unit: scores on a scale] — Fagerström test is a screening for alcohol consumption. This score ranges from 0 (Not/Very low dependency) to 10 (Very high dependency). Population: In smokers only (N=54)
  scores on a scale
    number analyzed (Participants) | 27 | 27 | 54
    (all) | 3.4 (2.6) | 3.4 (2.6) | 3.4 (2.6)
MADRS Score (Quantitative variable) [Mean (Standard Deviation); unit: scores on a scale] — MADRS (Montgomery and Asberg Depression Rating Scale) range from 0 (Normothymic) to 60 (medium depression).
  scores on a scale | 7.9 (7.6) | 7.9 (6.3) | 7.9 (6.9)
MADRS Score (Categorical variable) [Count of Participants; unit: Participants] — MADRS (Montgomery and Asberg Depression Rating Scale) range from 0 (Normothymic) to 60 (medium depression).
  Participants
    Normothymic | 30 | 28 | 58
    Mild depression | 15 | 21 | 36
    Depression Medium | 6 | 4 | 10
Score of Hamilton [Mean (Standard Deviation); unit: scores on a scale] — The Hamilton Depression Scale is a test for assessing the intensity of depressive symptoms. It ranges from 0 to 56. The higher the score is, the more severe the depression is.
  scores on a scale | 5.6 (6.1) | 5.6 (7.0) | 5.6 (6.5)
HEIQ (health Education Impact Questionnaire) score [Mean (Standard Deviation); unit: scores on a scale] — HEIQ (Health Education Impact Questionnaire) assesses the concept of empowerment (health-promoting behaviours, commitment, social integration, etc.).
  Its scores range from 0 to 160. Higher scores mean a better health-related empowerment .
  scores on a scale | 118.6 (11.7) | 118.6 (12.6) | 118.6 (12.1)
Standardised Quality of Life Scores (EORTC - QLQ-C30) [Mean (Full Range); unit: Standardized scores on a scale] — Standardised QLQ-C30 scoring according to EORTC scoring manual (Fayers et al. EORTC QLQ-C30 scoring manual. 2001).
  15 dimensions are presented below. Each dimension is a standardised score ranges from 0 to 100. A low score corresponds to a low functional level, an absence of symptoms or a low level of QoL/ overall health and, conversely, so that a high score corresponds to a high functional level, a high presence of symptoms or a high level of QoL/overall health. Population: Patients with available quality of life score
  Standardized scores on a scale
    Physical functioning: number analyzed (Participants) | 49 | 51 | 100
    Physical functioning | 80.8 [20.0 to 100.0] | 83.5 [46.7 to 100.0] | 82.2 [20.0 to 100.0]
    Role functioning: number analyzed (Participants) | 49 | 51 | 100
    Role functioning | 81.3 [16.7 to 100.0] | 80.1 [16.7 to 100.0] | 80.7 [16.7 to 100.0]
    Emotional functioning: number analyzed (Participants) | 49 | 51 | 100
    Emotional functioning | 74.9 [0.0 to 100.0] | 76.5 [0.0 to 100.0] | 75.7 [0.0 to 100.0]
    Cognitive functioning: number analyzed (Participants) | 49 | 51 | 100
    Cognitive functioning | 79.9 [0.0 to 100.0] | 77.8 [0.0 to 100.0] | 78.8 [0.0 to 100.0]
    Social functioning: number analyzed (Participants) | 49 | 51 | 100
    Social functioning | 76.2 [0.0 to 100.0] | 74.8 [0.0 to 100.0] | 75.5 [0.0 to 100.0]
    Fatigue: number analyzed (Participants) | 49 | 51 | 100
    Fatigue | 45.4 [0.0 to 100.0] | 42 [0.0 to 100.0] | 43.7 [0.0 to 100.0]
    Nausea and vomiting: number analyzed (Participants) | 49 | 51 | 100
    Nausea and vomiting | 8.5 [0.0 to 100.0] | 7.8 [0.0 to 50.0] | 8.2 [0.0 to 100.0]
    Pain: number analyzed (Participants) | 49 | 51 | 100
    Pain | 26.9 [0.0 to 100.0] | 23.9 [0.0 to 100.0] | 25.3 [0.0 to 100.0]
    Dyspnoea: number analyzed (Participants) | 49 | 51 | 100
    Dyspnoea | 24.5 [0.0 to 100.0] | 20.9 [0.0 to 100.0] | 22.7 [0.0 to 100.0]
    Insomnia: number analyzed (Participants) | 49 | 51 | 100
    Insomnia | 33.3 [0.0 to 100.0] | 34.0 [0.0 to 100.0] | 33.7 [0.0 to 100.0]
    Appetite loss: number analyzed (Participants) | 48 | 51 | 99
    Appetite loss | 15.3 [0.0 to 100.0] | 17.0 [0.0 to 100.0] | 16.2 [0.0 to 100.0]
    Constipation: number analyzed (Participants) | 49 | 51 | 100
    Constipation | 14.3 [0.0 to 100.0] | 15.7 [0.0 to 100.0] | 15.0 [0.0 to 100.0]
    Diarrhoea: number analyzed (Participants) | 49 | 51 | 100
    Diarrhoea | 10.2 [0.0 to 66.7] | 18.3 [0.0 to 100.0] | 14.3 [0.0 to 100.0]
    Financial difficulties: number analyzed (Participants) | 48 | 51 | 99
    Financial difficulties | 20.8 [0.0 to 100.0] | 25.5 [0.0 to 100.0] | 23.2 [0.0 to 100.0]
    Global health status/QoL (revised): number analyzed (Participants) | 48 | 51 | 99
    Global health status/QoL (revised) | 61.6 [0.0 to 100.0] | 65.4 [16.7 to 100.0] | 63.6 [0.0 to 100.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Individual Decrease of Tobacco Consumption at 3 Months
Description: Individual decrease of 20% in the AUDIT (Alcohol Use Disorders Identification Test) score observed at 3 months
  AUDIT test measures alcohol consumption and makes it possible to describe its profiles. Its score ranges from 0 (no consumption) to 28 (alcohol dependence).
Time Frame: 3 months
Population: Only patients with available data at 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 48 | 53
Participants
  Success | 23 | 19
  Success not maintained | 18 | 29
  Missing | 7 | 5

2. Primary Outcome: Number of Patients With Individual Decrease of Tobacco Consumption at 3 Months and Maintained at 6 Months
Description: Individual decrease of 20% in the AUDIT score observed at 3 months compared to the value collected at baseline and maintained at 6 months.
  Success depends on tobacco consumption at 3 months and 6 months.
  AUDIT test measures alcohol consumption and makes it possible to describe its profiles. Its score ranges from 0 to 28. Its score ranges from 0 (no consumption) to 28 (alcohol dependence).
Time Frame: 3 months and 6 months
Population: Only patients with available data at 3 months and 6 months
Measure: Number; unit: participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 48 | 53
participants
  Success | 17 | 14
  Success not maintained | 1 | 1
  Missing | 5 | 4

3. Secondary Outcome: Number of Patients With Individual Decreased of Alcohol and/or Tobacco Consumption
Description: Individual reduction of around 20% in the average daily consumption of alcohol and/or tobacco (calculated on the basis of consumption schedules) between inclusion and the first follow-up at 3 months (with no increase in the other consumption if the subject has both alcohol and tobacco consumption at inclusion).
Time Frame: 3 months
Population: Patients with tobacco or alcohol consumption at baseline and available data at 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 48 | 53
Participants
  Success | 12 | 15
  Failure | 22 | 26
  Missing | 14 | 12

4. Secondary Outcome: Number of Patients With Decreased Alcohol and/or Tobacco Consumption
Description: Individual reduction of around 20% in the average daily consumption of alcohol and/or tobacco (calculated on the basis of consumption schedules) between inclusion and the first follow-up at 3 months and a continuation of this reduction at the second follow-up at 6 months (with no increase in the other consumption if the subject has both alcohol and tobacco consumption at inclusion).
  Success depends on alcohol and tobacco level consumption at 3 months and 6 months.
Time Frame: 3 months and 6 months
Population: Patients with tobacco or alcohol consumption at baseline and data available at 3 months and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 12 | 15
Participants
  Success | 6 | 6
  Failure | 2 | 2
  Missing | 4 | 7

5. Secondary Outcome: Number of Patients Per Current Treatments at Baseline
Time Frame: Baseline
Population: Only patients with available data at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 51 | 53
Participants
  Surgery: Missing | 0 | 0
  Surgery: No | 50 | 52
  Surgery: Yes | 1 | 1
  Chemotherapy: Missing | 0 | 0
  Chemotherapy: No | 4 | 2
  Chemotherapy: Yes | 47 | 51
  Radiotherapy: Missing | 0 | 0
  Radiotherapy: No | 50 | 53
  Radiotherapy: Yes | 1 | 0
  Hormonotherapy: Missing | 0 | 0
  Hormonotherapy: No | 49 | 52
  Hormonotherapy: Yes | 2 | 1
  No treatment: Missing | 0 | 0
  No treatment: No | 51 | 52
  No treatment: Yes | 0 | 1

6. Secondary Outcome: Number of Patients Per Current Treatments at 3 Months
Time Frame: 3 months
Population: Only patients with available data at 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 51 | 53
Participants
  Surgery: Missing | 5 | 4
  Surgery: No | 40 | 47
  Surgery: Yes | 6 | 2
  Chemotherapy: Missing | 5 | 4
  Chemotherapy: No | 32 | 40
  Chemotherapy: Yes | 14 | 9
  Radiotherapy: Missing | 5 | 4
  Radiotherapy: No | 36 | 30
  Radiotherapy: Yes | 10 | 19
  Hormonotherapy: Missing | 5 | 4
  Hormonotherapy: No | 33 | 39
  Hormonotherapy: Yes | 13 | 10
  No treatment: Missing | 5 | 4
  No treatment: No | 36 | 36
  No treatment: Yes | 10 | 13

7. Secondary Outcome: Number of Patients Per Current Treatments at 6 Months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 51 | 53
Participants
  Surgery: Missing | 0 | 0
  Surgery: No | 49 | 53
  Surgery: Yes | 2 | 0
  Chemotherapy: Missing | 0 | 0
  Chemotherapy: No | 46 | 47
  Chemotherapy: Yes | 5 | 6
  Radiotherapy: Missing | 0 | 0
  Radiotherapy: No | 44 | 45
  Radiotherapy: Yes | 7 | 8
  Hormonotherapy: Missing | 0 | 0
  Hormonotherapy: No | 35 | 28
  Hormonotherapy: Yes | 16 | 25
  No treatment: Missing | 0 | 0
  No treatment: No | 42 | 43
  No treatment: Yes | 9 | 10

8. Secondary Outcome: Number of Patients Who Continued Psychotropic Treatment(s) at Baseline, 3 Months and 6 Months
Description: Ongoing psychotropic treatment(s) at baseline, 3 months and 6 months.
Time Frame: Baseline, 3 months and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 51 | 53
Participants
  Baseline: No | 35 | 35
  Baseline: Yes | 16 | 18
  Baseline: Missing | 0 | 0
  3 months: No | 34 | 35
  3 months: Yes | 12 | 14
  3 months: Missing | 5 | 4
  6 months: No | 29 | 30
  6 months: Yes | 8 | 14
  6 months: Missing | 14 | 9

9. Secondary Outcome: Number of Patients Who Has Current Monitoring With Regard to Behaviour/Emotional State
Description: Current monitoring with regard to behaviour/emotional state
Time Frame: Baseline, 3 months and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 51 | 53
Participants
  Baseline: Missing | 0 | 1
  Baseline: No | 38 | 36
  Baseline: Yes | 13 | 16
  3 months: Missing | 5 | 4
  3 months: No | 31 | 41
  3 months: Yes | 15 | 8
  6 months: Missing | 14 | 10
  6 months: No | 29 | 37
  6 months: Yes | 8 | 6

10. Secondary Outcome: Number of Patients Who by Type of Professional Monitored for Behaviour/Emotional State at Baseline
Description: Type of professional followed for behaviour/emotional state at baseline
Time Frame: Baseline
Population: Patients with current monitoring with regard to behaviour/emotional state
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 13 | 16
Participants
  Psychologist: No | 3 | 3
  Psychologist: Yes | 10 | 13
  Psychiatrist: No | 11 | 14
  Psychiatrist: Yes | 2 | 2
  Health professional specialising in tobaccoology and addiction: No | 13 | 15
  Health professional specialising in tobaccoology and addiction: Yes | 0 | 1
  Other professional: No | 12 | 16
  Other professional: Yes | 1 | 0

11. Secondary Outcome: Number of Patients Who by Type of Professional Monitored for Behaviour/Emotional State at 3 Months
Description: Type of professional followed for behaviour/emotional state at 3 months
Time Frame: 3 months
Population: Patients with current monitoring with regard to behaviour/emotional state
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 15 | 8
Participants
  Psychologist: No | 4 | 3
  Psychologist: Yes | 11 | 5
  Psychiatrist: No | 13 | 5
  Psychiatrist: Yes | 2 | 3
  Health professional specialising in tobaccoology and addiction: No | 15 | 8
  Health professional specialising in tobaccoology and addiction: Yes | 0 | 0
  Other professional: No | 13 | 8
  Other professional: Yes | 2 | 0

12. Secondary Outcome: Number of Patients by Type of Professional Monitored for Behaviour/Emotional State at 6 Months
Description: Type of professional followed for behaviour/emotional state at 6 months
Time Frame: 6 months
Population: Patients with current monitoring with regard to behaviour/emotional state
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 8 | 6
Participants
  Psychologist: No | 1 | 3
  Psychologist: Yes | 7 | 3
  Psychiatrist: No | 5 | 2
  Psychiatrist: Yes | 3 | 4
  Health professional specialising in tobaccoology and addiction: No | 7 | 6
  Health professional specialising in tobaccoology and addiction: Yes | 1 | 0
  Other professional: No | 8 | 6
  Other professional: Yes | 0 | 0

13. Secondary Outcome: AUDIT Score at Baseline, 3 Months, and 6 Months
Description: Alcohol Use Disorders Identification Test-Consumption (AUDIT-C) score ranges from 0 (No alcohol consumption) to 12 (alcohol dependence). Consumption profiles can be derived from this.
  Higher scores indicate a worse outcome: alcohol dependence.
Time Frame: Baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Arm 1: Arm 1 : Motivational Intervention group
  Motivational Intervention group: Participants in the intervention group a one-session brief motivational intervention administered by a psychologist. This intervention consist in a single adapted motivational interview lasting 20-30 minutes, based on the principles of the trans-theoretical model and on the manual for motivational therapy. It is carried out by the same psychologist, trained and supervised for this type of intervention.
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 51 | 53
score on a scale
  Baseline | 3.4 (4.2) | 2.9 (2.0)
  3 months | 3.6 (5.4) | 2.6 (1.8)
  6 months | 3.0 (4.9) | 2.7 (2.6)

14. Secondary Outcome: Currently, How Many Cigarettes Per Day do You Smoke on Average?
Time Frame: Baseline, 3 months and 6 months
Population: Only smokers who have completed form at baseline, 3 months and 6 months.
Measure: Mean (Standard Deviation); unit: Cigarettes per day
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 27 | 27
Cigarettes per day
  Baseline | 11.5 (8.1) | 10.8 (6.9)
  3 months: number analyzed (Participants) | 20 | 17
  3 months | 9.3 (6.1) | 10.4 (7.0)
  6 months: number analyzed (Participants) | 17 | 13
  6 months | 9.1 (6.9) | 11.0 (8.7)

15. Secondary Outcome: Number of Patients Who Consume Electronic Cigarettes
Time Frame: Baseline, 3 months and 6 months
Population: Only smokers at baseline (N=54), 3 months (N=37) and 6 months (N=30).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 27 | 27
Participants
  Baseline: No | 25 | 24
  Baseline: Yes | 2 | 3
  3 months: number analyzed (Participants) | 20 | 17
  3 months: No | 17 | 16
  3 months: Yes | 3 | 1
  6 months: number analyzed (Participants) | 17 | 13
  6 months: No | 15 | 12
  6 months: Yes | 2 | 1

16. Secondary Outcome: Type of Consumption of Electronic Cigarettes
Time Frame: Baseline, 3 months and 6 months
Population: Patient with electronic cigarette use and who answered the form
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 3 | 3
Participants
  Baseline: number analyzed (Participants) | 2 | 3
  Baseline: With nicotine | 1 | 3
  Baseline: Without nicotine | 1 | 0
  3 months: number analyzed (Participants) | 3 | 1
  3 months: With nicotine | 2 | 1
  3 months: Without nicotine | 1 | 0
  6 months: number analyzed (Participants) | 2 | 1
  6 months: With nicotine | 1 | 1
  6 months: Without nicotine | 1 | 0

17. Secondary Outcome: Fagerström Score
Description: Fagerström test assesses tobacco consumption and makes it possible to describe patterns of tobacco addiction. Its score ranges from 0 (non-addiction to smoking) to 10 (strong or very strong dependence on tobacco).
Time Frame: Baseline, 3 months, 6 months
Population: In smokers only (N=54 smokers at baseline)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 27 | 27
score on a scale
  Baseline | 3.4 (2.6) | 3.4 (2.6)
  3 months: number analyzed (Participants) | 20 | 17
  3 months | 3.7 (2.5) | 3.8 (2.1)
  6 months: number analyzed (Participants) | 17 | 13
  6 months | 3.0 (2.3) | 3.7 (2.7)

18. Secondary Outcome: MADRS Score
Description: MADRS (Montgomery-Åsberg Depression Rating Scale) assesses the severity of depression in patients with mood disorders. Its score ranges from 0 (normothymic) to 60 (depression).
Time Frame: Baseline, 3 months, 6 months
Population: Eligible and assessable patients who have completed the MADRS questionnaire at baseline, 3 months and 6 months. For this questionnaire, there were no missing data at each time point (baseline, 3 months and 6 months).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 51 | 53
score on a scale
  Baseline | 7.9 (7.6) | 7.9 (6.3)
  3 months | 8.5 (7.2) | 6.3 (5.8)
  6 months | 7.9 (7.9) | 4.8 (5.2)

19. Secondary Outcome: Score of Hamilton
Description: Hamilton test assesses symptoms of anxiety. Its score ranges from 0 to 56. The higher the score is, the more severe the depression is.
Time Frame: Baseline, 3 months and 6 months
Population: Eligible and assessable patients who have completed the Hamilton questionnaire at baseline, 3 months and 6 months. For this questionnaire, there were no missing data at each time point (baseline, 3 months and 6 months).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 51 | 53
score on a scale
  Baseline | 5.6 (6.1) | 5.6 (7.0)
  3 months | 4.5 (5.3) | 3.5 (4.1)
  6 months | 4.4 (6.0) | 2.6 (3.3)

20. Secondary Outcome: Standardised Quality of Life Scores (EORTC - QLQ-C30)
Description: QLQ-C30 questionnaire (EORTC) assesses quality of life across 15 dimensions :
  * 5 functional dimensions : Physical functioning, Role functioning, Emotional, Cognitive functioning, Social functioning;
  * 9 symptomatic dimensions: Fatigue, Nausea and vomiting, Pain, Dyspnea, Insomnia, Appetite loss, Diarrhoea, Financial difficulties;
  * 1 global health dimension: Global health status/QoL
  Each dimension is a standardised score ranges from 0 to 100. A low score corresponds to a low functional level, an absence of symptoms or a low level of QoL/ overall health and, conversely, so that a high score corresponds to a high functional level, a high presence of symptoms or a high level of QoL/overall health.
Time Frame: 3 months
Population: Participants who completed at least one item of the questionnaire. Note that some participants may not have completed the 30 items of the questionnaires, which explains why the number of participants differs for the different items of the questionnaires.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 51 | 53
scores on a scale
  Physical functioning: number analyzed (Participants) | 41 | 53
  Physical functioning | 81.0 (16.4) | 82.1 (18.1)
  Role functioning: number analyzed (Participants) | 41 | 53
  Role functioning | 84.6 (18.0) | 89.0 (17.8)
  Emotional functioning | 67.9 (27.0) | 76.3 (20.2)
  Cognitive functioning | 75.8 (27.1) | 81.6 (18.5)
  Social functioning | 70.6 (29.9) | 78.7 (24.3)
  Fatigue: number analyzed (Participants) | 41 | 53
  Fatigue | 42.0 (26.4) | 39.0 (21.1)
  Nausea and vomiting: number analyzed (Participants) | 41 | 53
  Nausea and vomiting | 5.3 (12.6) | 3.9 (7.9)
  Pain: number analyzed (Participants) | 41 | 53
  Pain | 26.4 (25.3) | 28.7 (21.3)
  Dyspnoea: number analyzed (Participants) | 41 | 53
  Dyspnoea | 15.4 (25.9) | 27.0 (19.2)
  Insomnia: number analyzed (Participants) | 41 | 53
  Insomnia | 42.3 (32.5) | 37.6 (30.8)
  Appetite loss: number analyzed (Participants) | 41 | 53
  Appetite loss | 14.6 (22.4) | 12.1 (18.9)
  Constipation: number analyzed (Participants) | 41 | 53
  Constipation | 8.9 (18.3) | 5.7 (12.7)
  Diarrhoea: number analyzed (Participants) | 41 | 46
  Diarrhoea | 4.9 (11.9) | 8.0 (22.4)
  Financial difficulties | 23.8 (32.3) | 21.3 (28.2)
  Global health status/QoL | 61.1 (17.9) | 64.2 (18.4)

21. Secondary Outcome: Standardised Quality of Life Scores (EORTC - QLQ-C30)
Description: as for outcome 20
Time Frame: 6 months
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 51 | 53
scores on a scale
  Physical functioning: number analyzed (Participants) | 37 | 41
  Physical functioning | 80.2 (18.5) | 86.0 (16.0)
  Role functioning: number analyzed (Participants) | 37 | 41
  Role functioning | 81.5 (24.1) | 88.2 (19.5)
  Emotional functioning: number analyzed (Participants) | 37 | 41
  Emotional functioning | 62.6 (28.7) | 75.6 (18.2)
  Cognitive functioning: number analyzed (Participants) | 37 | 41
  Cognitive functioning | 72.5 (30.2) | 78.5 (21.8)
  Social functioning: number analyzed (Participants) | 37 | 41
  Social functioning | 70.7 (33.4) | 81.7 (27.6)
  Fatigue: number analyzed (Participants) | 37 | 41
  Fatigue | 44.1 (23.6) | 31.4 (20.5)
  Nausea and vomiting: number analyzed (Participants) | 37 | 41
  Nausea and vomiting | 7.2 (20.6) | 4.1 (12.2)
  Pain: number analyzed (Participants) | 37 | 41
  Pain | 27.0 (27.0) | 26.8 (25.8)
  Dyspnoea: number analyzed (Participants) | 37 | 41
  Dyspnoea | 17.1 (24.4) | 21.1 (27.6)
  Insomnia: number analyzed (Participants) | 37 | 41
  Insomnia | 48.6 (33.0) | 37.4 (32.7)
  Appetite loss: number analyzed (Participants) | 37 | 41
  Appetite loss | 13.5 (24.2) | 3.3 (10.0)
  Constipation: number analyzed (Participants) | 37 | 41
  Constipation | 20.7 (31.8) | 9.8 (22.7)
  Diarrhoea: number analyzed (Participants) | 37 | 40
  Diarrhoea | 5.4 (18.4) | 7.5 (16.0)
  Financial difficulties: number analyzed (Participants) | 36 | 41
  Financial difficulties | 23.1 (33.6) | 22.8 (35.3)
  Global health status/QoL: number analyzed (Participants) | 37 | 41
  Global health status/QoL | 58.3 (20.7) | 63.6 (20.6)

22. Secondary Outcome: HEIQ Score
Description: HEIQ (Health Education Impact Questionnaire) assesses the concept of empowerment (health-promoting behaviours, commitment, social integration, etc.). Its scores range from 0 to 160. Higher scores mean a better health-related empowerment .
Time Frame: Baseline, 3 months, 6 months
Population: Patients with available score at baseline or 3 months or 6 months.
Measure: Median (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 51 | 53
scores on a scale
  Baseline | 119 (11.7) | 119 (12.6)
  3 months | 114 (11.2) | 117.5 (12.5)
  6 months | 118 (13.4) | 120 (12.5)

23. Secondary Outcome: Motivation Score to Change Consumption Habits (Alcohol/Tobacco)
Description: This score ranges from 0 to 140.
  The questionnaire consists of 14 questions on motivation to change alcohol/tobacco consumption habits, each with a response scale ranging from 0 (probably not) to 10 (probably).
  For each question, a sub-score ranges from 0 to 10 is given and then a total score of motivation to change consumption habits is calculated by adding up all the answers to the 14 items.
  The higher the score is, greater the patient's willingness to change his or her alcohol/tobacco consumption.
Time Frame: Baseline, 3 months and 6 months
Population: Patients with available score.
Measure: Median (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 51 | 53
scores on a scale
  Baseline | 121 (22.9) | 117.5 (32.0)
  3 months | 129 (29.0) | 126 (38.5)
  6 months | 120 (19.6) | 126 (31.7)

24. Secondary Outcome: Satisfaction Questionnaire
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 51 | 53
Participants
  Do you think it would be important to ask cancer patients about their consumption behaviour?: Missing | 14 | 6
  Do you think it would be important to ask cancer patients about their consumption behaviour?: No | 1 | 2
  Do you think it would be important to ask cancer patients about their consumption behaviour?: Yes | 30 | 42
  Do you think it would be important to ask cancer patients about their consumption behaviour?: Don't know | 6 | 3
  Would it be useful to ask cancer patients about their alcohol/tobacco consumption behaviour: Missing | 14 | 7
  Would it be useful to ask cancer patients about their alcohol/tobacco consumption behaviour: No | 1 | 1
  Would it be useful to ask cancer patients about their alcohol/tobacco consumption behaviour: Yes | 33 | 40
  Would it be useful to ask cancer patients about their alcohol/tobacco consumption behaviour: Don't know | 3 | 5
  Would you have liked the questions on consumption to have been asked at another time?: Missing | 16 | 6
  Would you have liked the questions on consumption to have been asked at another time?: No | 29 | 41
  Would you have liked the questions on consumption to have been asked at another time?: Yes | 6 | 6
  Would you have liked the questions on consumption to have been asked at another time?: Don't know | 0 | 0

25. Secondary Outcome: On a Scale of 1 to 10 How Would You Rate Your Overall Satisfaction With Having Benefited From a Brief Intervention at the Bergonié Institute?
Description: Satisfaction score ranges from 1 to 10. Low scores indicate less satisfaction.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 51 | 53
Participants
  Missing | 15 | 6
  3 | 0 | 1
  5 | 3 | 5
  6 | 2 | 4
  7 | 0 | 3
  8 | 11 | 17
  9 | 8 | 6
  10 | 12 | 11

ADVERSE EVENTS:
Time Frame: Adverse events were not collected for this study.
Description: Adverse events were not collected for this study.
Arm/Group | Groupe 1 | Groupe 2
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2015-10-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT03371732/Prot_000.pdf